CLINICAL TRIAL: NCT03866187
Title: A first-time-in Human (FTIH), Phase I/II, Randomized, Multi-centric, Single-blind, Controlled Dose-escalation Study to Evaluate the Reactogenicity, Safety, Immunogenicity and Efficacy of GSK Biologicals' HBV Viral Vector Vaccines Given in a Prime-boost Schedule With Sequential or Co-administration of Adjuvanted Proteins Therapeutic Vaccine (GSK3528869A) in Chronic Hepatitis B Patients (18-65 Years Old) Well Controlled Under Nucleo(s)Tide Analogue (NA) Therapy
Brief Title: Safety, Efficacy, Immunogenicity Study of GSK Biologicals' HBV Viral Vector and Adjuvanted Proteins Vaccine (GSK3528869A) in Adult Patients With Chronic Hepatitis B Infection
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Following the primary phase(24 weeks post last vaccination)the predefined efficacy endpoint was not met.Noting the lack of efficacy and with the objective to prioritize patients'safety GSK has decided on the early termination of the study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 204852; 2017-001452-55 (EudraCT Number)
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: Study will be conducted following a staggered design overseen by Internal Safety Review Committee (iSCR):
  * Step A (low dose of each vaccine): Approximately 15 patients will be randomized (1:1:1). Fourteen days after the 2nd vaccination, iSRC will review all available safety data (of at least 12 patients if approved by local authorities). If considered appropriate to continue, Step B will start.
  * Step B (prime-boost with ChAd155-hIi-HBV and Modified Vaccinia Ankara HBV vaccine (MVA-HBV) and sequential administration with HBc-HBs/AS01B-4): Approximately 40 patients will first be randomized (2:1:1) for vaccination. Fourteen days after the 2nd vaccination, iSRC will review all available safety data. If considered appropriate to continue, approximately 36 additional patients will be randomized for vaccination.
  * Step C (prime-boost with ChAd155-hIi-HBV and MVA-HBV and co-administration with HBc-HBs/AS01B-4): Step C randomization (2:1) will start post completion of Step B enrolment.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group A1_Step A (Experimental): Subjects aged 18-65 years receive one dose of each of the study vaccines, Chimpanzee adenovirus HBV vaccine (ChAd155-hIi-HBV) low dose formulation at Day 1, Modified Vaccinia Ankara HBV vaccine (MVA-HBV) low dose formulation at Day 57 and two doses of HBc-HBs/AS01B-4 low dose formulation, one at Day 113 and one at Day 169.
  Interventions: Biological: ChAd155-hIi-HBV low dose formulation; Biological: HBc-HBs/AS01B-4 low dose formulation; Biological: MVA-HBV low dose formulation
- Group A2_Step A (Active Comparator): Subjects aged 18-65 years receive four doses of the study vaccine HBc-HBs/AS01B-4 low dose formulation, one dose each at Days 1, 57, 113 and 169.
  Interventions: Biological: HBc-HBs/AS01B-4 low dose formulation
- Group A3_Step A (Placebo Comparator): Subjects aged 18-65 years receive four doses of placebo, one dose each at Days 1, 57, 113 and 169.
  Interventions: Drug: Placebo
- Group B1_Step B (Experimental): Subjects aged 18-65 years receive one dose of each of the study vaccines, ChAd155-hIi-HBV high dose formulation at Day 1, MVA-HBV high dose formulation at Day 57 and two doses of HBc-HBs/AS01B-4 high dose formulation, one at Day 113 and one at Day 169.
  Interventions: Biological: ChAd155-hIi-HBV high dose formulation; Biological: HBc-HBs/AS01B-4 high dose formulation; Biological: MVA-HBV high dose formulation
- Group B2_Step B (Active Comparator): Subjects aged 18-65 years receive four doses of the study vaccine HBc-HBs/AS01B-4 high dose formulation, one dose each at Days 1, 57, 113 and 169.
  Interventions: Biological: HBc-HBs/AS01B-4 high dose formulation
- Group B3_Step B (Active Comparator): Subjects aged 18-65 years receive two doses of placebo, one each at Days 1 and 57, one dose of ChAd155-hIi-HBV high dose formulation at Day 113 and one dose of MVA-HBV high dose formulation at Day 169.
  Interventions: Biological: ChAd155-hIi-HBV high dose formulation; Biological: MVA-HBV high dose formulation; Drug: Placebo
- Group C1_Step C (Experimental): Subjects aged 18-65 years receive one dose of ChAd155-hIi-HBV high dose formulation co-administered with HBc-HBs/AS01B-4 high dose formulation at Day 1 and the 3 following doses of MVA-HBV high dose formulation co-administered with HBc-HBc-HBs/AS01B-4 high dose formulation at Day 57, 113 and Day 169.
  Interventions: Biological: ChAd155-hIi-HBV high dose formulation; Biological: HBc-HBs/AS01B-4 high dose formulation; Biological: MVA-HBV high dose formulation
- Group C2_Step C (Active Comparator): Subjects aged 18-65 years receive two doses of placebo at Days 1 and 57, one dose of ChAd155-hIi-HBV high dose formulation co-administered with HBc-HBs/AS01B-4 high dose formulation at Day 113 and one dose of MVA-HBV high dose formulation co-administered with HBc-HBs/AS01B-4 high dose formulation at Day 169.
  Interventions: Biological: ChAd155-hIi-HBV high dose formulation; Biological: HBc-HBs/AS01B-4 high dose formulation; Biological: MVA-HBV high dose formulation; Drug: Placebo

INTERVENTIONS:
Biological: ChAd155-hIi-HBV low dose formulation — Subjects in group A1 receive one dose of ChAd155-hIi-HBV low dose formulation at Day 1, by intramuscular injection in the deltoid of the non-dominant arm.
  Arms: Group A1_Step A
Biological: ChAd155-hIi-HBV high dose formulation — Subjects in groups B1 and B3 receive one dose of ChAd155-hIi-HBV high dose formulation at Day 1 and Day 113 respectively, by intramuscular injection in the deltoid of the non-dominant arm.
  Subjects in groups C1 and C2 receive one dose of ChAd155-hIi-HBV high dose formulation at Day 1 and Day 113 respectively, by intramuscular injection in the deltoid of the dominant arm.
  Arms: Group B1_Step B; Group B3_Step B; Group C1_Step C; Group C2_Step C
Biological: HBc-HBs/AS01B-4 low dose formulation — Subjects in group A1 receive two doses of HBc-HBs/AS01B-4 low dose formulation, one at Day 113 and one at Day 169 and subjects in group A2 receive four doses of the low dose formulation, one dose each at Days 1, 57, 113 and 169, by intramuscular injection in the deltoid of the non-dominant arm.
  Arms: Group A1_Step A; Group A2_Step A
Biological: HBc-HBs/AS01B-4 high dose formulation — Subjects in group B1 receive two doses of HBc-HBs/AS01B-4 high dose formulation, one at Day 113 and one at 169; subjects in group B2 receive four doses, one dose each at Days 1, 57, 113 and 169; subjects in group C1 receive four co-administered doses at Days 1, 57, 113 and 169 and subjects in group C2 receive two co-administered doses at Days 113 and 169, by intramuscular injection in the deltoid of the non-dominant arm.
  Arms: Group B1_Step B; Group B2_Step B; Group C1_Step C; Group C2_Step C
Biological: MVA-HBV low dose formulation — Subjects in group A1 receive one dose of MVA-HBV low dose formulation at Day 57, by intramuscular injection in the deltoid of the non-dominant arm.
  Arms: Group A1_Step A
Biological: MVA-HBV high dose formulation — Subjects in groups B1 and B3 receive one dose of MVA-HBV high dose formulation at Day 57 and Day 169 respectively, by intramuscular injection in the deltoid of the non-dominant arm.
  Subjects in group C1 receive three co-administered doses of the vaccine at Days 57, 113 and 169 and subjects in group C2 receive one co-administered dose of the vaccine at Day 169, by intramuscular injection in the deltoid of the dominant arm.
  Arms: Group B1_Step B; Group B3_Step B; Group C1_Step C; Group C2_Step C
Drug: Placebo — Subjects in group A3 receive four doses of placebo, one each at Days 1, 57, 113 and 169 and subjects in group B3 receive two doses of placebo one each at Days 1 and 57, by intramuscular injection in the deltoid of the non-dominant arm. Subjects in group C2 receive 2 co-administered doses of placebo at Days 1 and 57, by intramuscular injection in the deltoid of the dominant and non-dominant arm.
  Arms: Group A3_Step A; Group B3_Step B; Group C2_Step C

SUMMARY:
A First-Time-In-Human study on GSK's therapeutic vaccines to evaluate the reactogenicity, safety, immunogenicity and efficacy on reduction of serum HBV surface antigen in HBV suppressed subjects under nucleo(s)tide treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the patient prior to performing any study specific procedure.
* A male or female between, and including, 18 and 65 years of age at the time of the first vaccination.
* Female patients of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as hysterectomy, bilateral ovariectomy or post-menopause.
* Female patients of childbearing potential may be enrolled in the study if the patient:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test at Screening, and
  * has agreed to continue adequate contraception from Screening until 12 weeks after completion of the vaccination series
* Male patients:

  * with documented bilateral vasectomy and resultant azoospermia, bilateral orchiectomy or azoospermia, or
  * who agree to practice abstinence from penile-vaginal intercourse (when this is their preferred and usual lifestyle) or use condoms from Screening until 12 weeks after completion of the vaccination series.
* Chronic Hepatitis B (CHB) patient, under and adherent to treatment with a nucleo(s)tide analogue with high barrier to resistance given as per approved label/dosage for at least 24 months.
* Documented medical history of Hepatitis B Virus e Antigen (HBeAg)-negative CHB prior to onset of NA therapy (applicable to all patients in Step A and Step B and to some patients in Step C) or documented medical history of HBeAg-negative CHB over a period of at least 24 months prior screening (applicable to some patients in Step C only).
* Documented HBV viral suppression as per local clinical diagnosis within the previous 24 months AND at Screening test HBV DNA < 10 IU/mL. If no results are available, two Screening tests need to be performed at least 2 weeks apart. Small fluctuations of HBV DNA (≤ 10 x LLOQ; LLOQ defined by laboratory that performed testing) are allowed provided HBV DNA is < 10 IU/mL at Screening and was clearly not rising during the previous 24 months.
* Documented normal level of ALT as per local clinical diagnosis within the previous 24 months AND at Screening test ALT < 48U/L. Small fluctuations of ALT (≤ 1.5 X ULN) are allowed provided ALT< 48 U/L at Screening. If no results are available, two Screening tests need to be performed at least 2 weeks apart. ULN are to be defined according to local laboratory reference range.
* No clinical diagnosis of cirrhosis (e.g. F4 by METAVIR scoring system or ≥ 6 by Ishak scoring system or FibroScan TE score > 12.5 kPa) within the previous 24 months.
* FibroScan Transient Elastography (TE) score < 9.6 kPa and FibroTest score < 0.59 at Screening. A patient with one of these parameters out of range, but having the liver biopsy within 12 months before screening that showed F0-2 by METAVIR scoring system or stage 0-4 by Ishak scoring system, can be included.
* HBsAg concentration > 50 IU/mL and anti-HBs negative at Screening.
* Anti-HBc positive at Screening.
* HBeAg-negative at Screening.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines during the period starting 30 days before the first dose of study vaccines, or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone ≥ 10 mg/day or equivalent. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the first dose of study vaccines or planned administration during the study period.
* Use of systemic cytotoxic agents, chronic antiviral agents or Chinese herbal medicines which, in the opinion of the investigator, may have activity against HBV within the previous 6 months prior to randomization into this study. Antiviral treatment/prevention for influenza or herpes simplex virus is allowed.
* Administration of adenovirus/adenovector-based or MVA-based vaccine within the last 12 months except for adenovirus/adenovector-based COVID-19 vaccines that could be administered up to 30 days prior to the first study vaccine dose (applicable for all patients except for the patients in France) OR Administration of adenovirus/adenovector-based or MVA-based vaccine within the last 12 months (applicable for the patients in France only).
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 14 days before each dose and ending 30 days after each dose of vaccines, with the exception of influenza vaccine that may be given at any time except within a 7-day period before or after each vaccine dose and COVID-19 vaccine that may be given at any time except within a 30-day period before or after each vaccine dose apart from COVID-19 mRNA based-vaccines that may be administered any time except for the period of 14 days before and 30 days after each study vaccine dose. Note: If the type of COVID-19 vaccine is unknown, the allowed interval of 30 days before or after each study vaccine dose should be followed.
* Treatment with nephrotoxic drugs or competitors of renal excretion within 2 months prior to Screening or the expectation that patient will receive any of these during the course of the study. TAF/TDF given as NA therapy is allowed.
* Concurrently participating in another clinical study, at any time during the study period, in which the patient has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Medical history of cirrhosis or hepatic decompensation.
* Planned for liver transplantation or previous liver transplantation.
* Personal or family (first degree) history of autoimmune disease.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Evidence of Hepatitis C Virus and hepatitis D Virus infection.
* Suspicion of or confirmed Hepatocellular Carcinoma or any other liver cancer in medical history or at Screening:

  * Suspicious foci at liver imaging exam
  * Elevated α-fetoprotein > 50 ng/mL.
* Documented evidence of other currently active cause of hepatitis.
* Hematology and biochemistry parameters outside normal clinical range at Screening:

Biochemistry:

* Glomerular filtration rate < 60 mL/min
* Bilirubin > 27.5 µmol/L unless *or the diagnosis of Gilbert Syndrome has been established and confirmed by the Investigator
* GGT > 65 U/L (males) or > 45 U/L (females)*
* ALT > 48 U/L
* AST > 42 U/L*
* ALP > 125 U/L*

Hematology:

* Hemoglobin < 12.0 g/dL (females) or < 13.5 g/dL (males)*
* Red blood cell count < 3.9 x 10^6 cells/mm^3 (females) or < 4.4 x 10^6 cells/mm^3 (males)*
* White blood cell count < 3,500 cells/mm^3 or > 12,000 cells/mm^3*
* Platelets < 140,000 cells/mm^3
* INR > 1.32 (i.e. 1.1 x ULN) *unless it is considered as clinically not significant by the Investigator

  * Known diabetes Type I.
  * Body Mass Index > 35 kg/m^2 at Screening.
  * Any serious or active medical or psychiatric illnesses other than chronic hepatitis B which, in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol.
  * History of or current drug abuse and/or excess of alcohol consumption as defined per local guidelines.
  * HIV-positive patient.
  * Pregnant or lactating female.
  * Female planning to become pregnant or planning to discontinue contraceptive precautions in the period starting from the Screening Visit up to 12 weeks post-last vaccination visit.
  * Fever and or acute minor illness may be enrolled for Screening at the discretion of the investigator, provided that the condition is resolved at the time of vaccination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting solicited local adverse events (AEs) | Within 7 days after each vaccination (from day of vaccination to 6 days after vaccination)
  The following local AEs are solicited: pain at injection site, redness at injection site and swelling at injection site.
Number of subjects reporting solicited general AEs | Within 7 days after each vaccination (from day of vaccination to 6 days after vaccination)
  The following general AEs are solicited: fatigue, fever*, gastrointestinal symptoms**, headache, myalgia and chills.
  *Fever is defined as temperature ≥38.0°C / 100.4°F. The preferred location for measuring temperature in this study is the oral cavity.
  **Gastrointestinal symptoms include nausea, vomiting, diarrhoea and/or abdominal pain.
Number of subjects reporting unsolicited AEs | Within 30 days after each vaccination (from day of vaccination to 29 days after vaccination)
  Unsolicited AE is defined as an AE reported in addition to those solicited during the clinical study and as any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Number of subjects with hematological, biochemical or urinalysis laboratory abnormalities | Within 30 days after each vaccination (from day of vaccination to 29 days after vaccination)
  Clinically significant abnormal laboratory findings (e.g. clinical chemistry, haematology, urinalysis) are reported.
  The investigator exercises his or her medical and scientific judgement in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant.
Number of subjects reporting serious adverse events (SAEs) | From Day 1 up to Day 337 (6 months after last dose)
  SAEs assessed include any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study patient.
Number of subjects reporting potential immune-mediated diseases (pIMDs) | From Day 1 up to Day 337 (six months after the last dose)
  pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Number of subjects reporting liver-disease-related (LDR) AEs | From Day 1 up to Day 337 (six months after the last dose)
  LDR AEs are defined as AEs related to the underlying chronic HBV infection and characterized by one or more of the following:
  Alanine Transaminase (ALT) flares
  * Elevation of ALT > 3 X Upper Limit of Normal (ULN):
    * Mild: > 3-5 X ULN
    * Moderate: > 5-10 X ULN
    * Severe: > 10 X ULN ALT flares with other substantial biochemical changes
  * Bilirubin ≥ 2 X ULN
  * And/or International Normalized Ratio (INR) > 1.5 Hepatic decompensation Occurrence of one or more of the following events: ascites, spontaneous bacterial peritonitis, hepatorenal syndrome, variceal bleeding, or hepatic encephalopathy.
  HBV-Deoxyribonucleic Acid (DNA) breakthrough Any increase in serum HBV DNA by >1 log10 from nadir or redetection of serum HBV DNA at levels 10-fold the Lower Limit of Quantification (LLOQ) of the viral load after HBV DNA was undetectable.
Number of subjects reporting any hematological adverse events of specific interest (AESIs) | From Day 1 up to Day 337 (six months after last dose)
  Hematological AESI is defined as:
  * Spontaneous local or general bleeding with thrombocytes < 50,000 platelets/mm^3
  * Anemia with hemoglobin < 9.5 g/dL.
Number of subjects reporting medically-attended adverse events (MAEs) | From Day 1 up to Day 337 (six months after the last dose)
  MAEs are defined as events for which the subject receives medical attention defined as hospitalization, or an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits.

SECONDARY OUTCOMES:
Number of seropositive subjects for anti-hepatitis B core antibody (anti-HBc) | At Days 1,15, 71, 113, 127, 183, 337, 505 and 841
  A seropositive subject is a subject whose antibody concentration is greater than or equal to the defined cut-off value.
Evaluation of immunogenicity in terms of Anti-HBc antibody concentration | At Days 1,15, 71, 113, 127, 183, 337, 505 and 841
  Antibody concentrations are presented as geometric mean concentrations (GMCs) of anti-HBc antibodies.
Number of subjects with anti-hepatitis B surface antigen (anti-HBs) seroconversion | At Days 1,15, 71, 113, 127, 183, 337, 505 and 841
  A seroconverted subject is a subject whose antibody concentration is above the lower limit of quantitation (LLOQ) of the assay.
Evaluation of immunogenicity in terms of anti-HBs antibody concentration | At Days 1,15, 71, 113, 127, 183, 337, 505 and 841
  Antibody concentrations are presented as geometric mean concentrations (GMCs) of anti-HBs antibodies.
Number of subjects with anti-HBs antibody concentration equal to or above 10 mIU/mL | At Days 1,15, 71, 113, 127, 183, 337, 505 and 841
  The number of subjects with anti-HBs antibody concentrations equal to or above 10 mIU/mL is reported.
Number of subjects with anti-HBs antibody concentration equal to or above 100 mIU/mL | At Days 1,15, 71, 113, 127, 183, 337, 505 and 841
  The number of subjects with anti-HBs antibody concentrations equal to or above 100 mIU/mL is reported.
Frequency of HBs-specific CD4+ T-cells | At Days 1,15, 57, 64, 71, 113, 127, 169, 183, 337, 505 and 841
  Frequency of HBs-specific CD4+ T-cells is expressed as HBs-specific CD4+ T-cells per million peripheral blood mononuclear cells (HBs-specific CD4+ T-cells/million PBMCs).
Frequency of HBs-specific CD8+ T-cells | At Days 1,15, 57, 64, 71, 113, 127, 169, 183, 337, 505 and 841
  Frequency of HBs-specific CD8+ T-cells is expressed as HBs-specific CD8+ T-cells per million peripheral blood mononuclear cells (HBs-specific CD8+ T-cells/million PBMCs).
Frequency of HBc-specific CD4+ T-cells | At Days 1,15, 57, 64, 71, 113, 127, 169, 183, 337, 505 and 841
  Frequency of HBc-specific CD4+ T-cells is expressed as HBc-specific CD4+ T-cells per million peripheral blood mononuclear cells (HBc-specific CD4+ T-cells/million PBMCs).
Frequency of HBc-specific CD8+ T-cells | At Days 1,15, 57, 64, 71, 113, 127, 169, 183, 337, 505 and 841
  Frequency of HBc-specific CD8+ T-cells is expressed as HBc-specific CD8+ T-cells per million peripheral blood mononuclear cells (HBc-specific CD8+ T-cells/million PBMCs).
Frequency of HBs-specific CD4+ T-cells responders | At Days 1,15, 57, 64, 71, 113, 127, 169, 183, 337, 505 and 841
  The number of HBs-specific CD4+ T-cells responders is reported.
Frequency of HBc-specific CD4+ T-cells responders | At Days 1,15, 57, 64, 71, 113, 127, 169, 183, 337, 505 and 841
  The number of HBc-specific CD4+ T-cells responders is reported.
Frequency of HBs-specific CD8+ T-cells responders | At Days 1,15, 57, 64, 71, 113, 127, 169, 183, 337, 505 and 841
  The number of HBs-specific CD8+ T-cells responders is reported.
Frequency of HBc-specific CD8+ T-cells responders | At Days 1,15, 57, 64, 71, 113, 127, 169, 183, 337, 505 and 841
  The number of HBc-specific CD8+ T-cells responders is reported.
Number of subjects with ≥ 0.5 log decrease of qHBsAg since pre-vaccination | At Days 1, 31, 57, 87, 113, 143, 169, 199, 225, 281, 337, 421, 505, 673, 841
  The number of subjects with ≥ 0.5 log decrease of qHBsAg since pre-vaccination is reported. Note: For study participants in Step B and Step C, Visits 19 (Day 253) and 21 (Day 309) are cancelled, which is why Day 253 and Day 309 time points are not reflected in the time frame.
Number of subjects with ≥ 1 log decrease of qHBsAg since pre-vaccination | At Days 1, 31, 57, 87, 113, 143, 169, 199, 225, 281, 337, 421, 505, 673, 841
  The number of subjects with ≥ 1 log decrease of qHBsAg since pre-vaccination is reported. Note: For study participants in Step B and Step C, Visits 19 (Day 253) and 21 (Day 309) are cancelled, which is why Day 253 and Day 309 time points are not reflected in the time frame.
Number of subjects with qHBsAg loss | At Days 1, 31, 57, 87, 113, 143, 169, 199, 225, 281, 337, 421, 505, 673, 841
  The number of subjects with qHBsAg loss since pre-vaccination is reported. Note: For study participants in Step B and Step C, Visits 19 (Day 253) and 21 (Day 309) are cancelled, which is why Day 253 and Day 309 time points are not reflected in the time frame.
Changes in qHBsAg since pre-vaccination | At Days 1, 31, 57, 87, 113, 143, 169, 199, 225, 281, 337, 421, 505, 673, 841
  Changes in serum qHBsAg since pre-vaccination are evaluated and expressed in log10 International Unit per milliliter (IU/mL). Note: For study participants in Step B and Step C, Visits 19 (Day 253) and 21 (Day 309) are cancelled, which is why Day 253 and Day 309 time points are not reflected in the time frame.
Number of subjects with HBsAg loss and anti-HBs seroconversion | At Days 1, 337, 505 and 841
  A subject is counted only when both HBsAg loss and anti-HBs seroconversion are reported for the subject.
  A seroconverted subject is a subject whose antibody concentration is above the LLOQ of the assay.
Evaluation of qHBsAg geometric mean concentrations | At Day 1, 31, 57, 87, 113, 143, 169, 199, 225, 281, 337, 421, 505, 673, 841
  The geometric mean of qHBsAg is reported. Note: For study participants in Step B and Step C, Visits 19 (Day 253) and 21 (Day 309) are cancelled, which is why Day 253 and Day 309 time points are not reflected in the time frame.
Number of subjects reporting any SAEs and SAEs causally related to an investigational vaccine | Throughout the study period (from Day 1 up to Day 841)
  SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study patient.
Number of subjects reporting MAEs | Throughout the study period (from Day 1 up to Day 841)
  MAEs are defined as events for which the subject receives medical attention defined as hospitalization, or an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits.
Number of subjects reporting pIMDs | Throughout the study period (from Day 1 up to Day 841)
  pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Number of subjects reporting liver-disease-related AEs | Throughout the study period (from Day 1 up to Day 841)
  LDR AEs are defined as AEs related to the underlying chronic HBV infection and characterized by one or more of the following:
  ALT flares
  • Elevation of ALT > 3 X ULN:
  * Mild: > 3-5 X ULN
  * Moderate: > 5-10 X ULN
  * Severe: > 10 X ULN
  ALT flares with other substantial biochemical changes
  * Bilirubin ≥ 2 X ULN
  * And/or INR > 1.5
  Hepatic decompensation Occurrence of one or more of the following events: ascites, spontaneous bacterial peritonitis, hepatorenal syndrome, variceal bleeding, or hepatic encephalopathy.
  HBV-DNA breakthrough Any increase in serum HBV DNA by >1 log10 from nadir or redetection of serum HBV DNA at levels 10-fold the LLOQ of the viral load after HBV DNA was undetectable.
Number of subjects reporting spontaneous local or general bleeding with thrombocytopenia | Throughout the study period (from Day 1 up to Day 841)
  Spontaneous local or general bleeding with thrombocytopenia defined as < 50,000 platelets/mm^3.
Number of subjects reporting anemia | Throughout the study period (from Day 1 up to Day 841)
  Anemia is defined as Hemoglobin < 9.5 g/dL.
Number of subjects reporting AEs and SAEs leading to study withdrawal | Throughout the study period (from Day 1 up to Day 841)
  The number of patients who experienced at least one AE or SAE leading to study withdrawal during the entire study period is reported.
Number of subjects reporting pregnancy and outcomes of reported pregnancy | Throughout the study period (from Day 1 up to Day 841)
  The number of patients who experienced pregnancy during the entire study period is to be reported, with pregnancy outcome.
  Pregnancy outcomes include:
  * Live infant NO apparent congenital anomaly
  * Live infant congenital anomaly
  * Stillbirth NO apparent congenital anomaly
  * Stillbirth congenital anomaly
  * Premature live infant NO apparent congenital anomaly
  * Premature live infant congenital anomaly
  * Spontaneous abortion NO apparent congenital anomaly
  * Spontaneous abortion congenital anomaly
  * Elective termination NO apparent congenital anomaly
  * Elective termination congenital anomaly
  * Therapeutic abortion
  * Ectopic pregnancy
  * Pregnancy ongoing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (37):
- Belgium (4):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
- France (4):
  - GSK Investigational Site, Clichy
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Strasbourg
- Germany (8):
  - GSK Investigational Site, Aachen
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bonn
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Tübingen
- GSK Investigational Site, Pokfulam, Hong Kong
- Poland (4):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Mysłowice
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Łańcut
- Spain (8):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
  - GSK Investigational Site, TorrejOn Ardoz Madrid
- Taiwan (4):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com